CLINICAL TRIAL: NCT02297529
Title: A Phase 3b, Multicenter, Open-label, Single-arm, Expanded Access Protocol of Talimogene Laherparepvec for the Treatment of Subjects in Europe With Unresected Stage IIIB to IVM1c Melanoma
Brief Title: Expanded Access Study of Talimogene Laherparepvec for Treatment of Subjects With Unresected Stage IIIB-IVM1c Melanoma
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120328; 2014-002834-30 (EudraCT Number)
Record Dates: First submitted 2014-10-17; First posted 2014-11-21 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Unresected Stage IIIB to IVM1c Melanoma
Keywords: unresected, Melanoma, expanded access, EU
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Open label single arm study. The initial dose of talimogene laherparepvec is up to 4.0 mL of 106 PFU/mL. Subsequent doses of talimogene laherparepvec are up to 4.0 mL of 108 PFU/mL.

SUMMARY:
The study is a phase 3b, multicenter, open-label, single-arm study designed to provide expanded access of Talimogene Laherparepvec for the treatment of subjects with unresected stage IIIB to IVM1c melanoma. The study will also evaluate the safety and tolerability of Talimogene Laherparepvec.

DETAILED DESCRIPTION:
This is a phase 3b, multicenter, open-label, single-arm, expanded access study of talimogene laherparepvec for the treatment of subjects with unresected stage IIIB to IVM1c melanoma in select European countries. Subjects with unresected stage lllB-IVM1c melanoma who are not eligible for or cannot access ongoing talimogene laherparepvec clinical trials and who meet the eligibility criteria outlined will be considered for participation in this protocol. Eligible subjects will be treated with talimogene laherparepvec until the subject has achieved a complete response, all injectable tumors have disappeared, clinically relevant (resulting in clinical deterioration or requiring change of therapy) disease progression beyond 6 months of therapy, intolerance of protocol treatment, or until talimogene laherparepvec receives marketing authorization approval in Europe for the treatment of melanoma, whichever occurs first. Subjects will be followed for safety approximately 30 (+7) days after the end of treatment. Thereafter, subjects who provide consent will be followed under an ongoing separate registry protocol for the long-term survival follow-up of subjects treated with talimogene laherparepvec in clinical trials. The registry protocol will also monitor for late and long-term adverse events thought to be potentially related to talimogene laherparepvec.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to initiation of any protocol-specific activities/procedures.
2. Male or female age ≥ 18 years at the time of informed consent.
3. Histologically confirmed diagnosis of melanoma
4. Subject has unresected stage lllB to IVM1c melanoma regardless of prior therapy
5. Subject who is not eligible for or cannot access ongoing talimogene laherparepvec clinical trials 6.Subject does not qualify for, or cannot access, other comparable or satisfactory alternative therapy for stage IIIB to IVM1c melanoma

7. Candidate for intralesional therapy 8. Adequate organ function. 9. ECOG performance status of 0, 1, or 2.

Exclusion Criteria:

1. Clinically active cerebral metastases.
2. Greater than 3 visceral metastases.
3. Bone metastases
4. Primary ocular or mucosal melanoma.
5. History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease.
6. Active herpetic skin lesions or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis)
7. Known to have acute or chronic active hepatitis B or C infection
8. Known to have human immunodeficiency virus infection
9. History of other malignancy within the past 3 years
10. Female subject is pregnant or breast-feeding, or planning to become pregnant during protocol treatment and through 3 months after the last dose of talimogene laherparepvec
11. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during protocol treatment and through 3 months after the last dose of talimogene laherparepvec.
12. Subject has known sensitivity to any of the products or components to be administered during dosing.
13. Subject has entered this protocol previously.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- Switzerland (3):
  - Research Site, Chur
  - Research Site, Lausanne
  - Research Site, Zurich

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com